CLINICAL TRIAL: NCT00589173
Title: An Interactive Preventive Health Record (IPHR) to Promote Patient-Centered Preventive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PD300045; RFA-07-007
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Prevention
Keywords: Preventive Care; Health information technology; Personal health record

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients referred to the IPHR
  Interventions: Behavioral: Interactive Preventive Health Record (IPHR)
- Control (Active Comparator): Patients receiving "standard" preventive care
  Interventions: Behavioral: "Standard" preventive care

INTERVENTIONS:
Behavioral: Interactive Preventive Health Record (IPHR) — Preventive health record designed to a) show patients the status of their preventive care recorded in their electronic record and b) make recommendations on what USPSTF endorsed preventive services that the user needs to receive.
  Arms: Intervention
Behavioral: "Standard" preventive care — Existing mechanisim for receiving preventive care in primary care (i.e. patients not referred to the IPHR).
  Arms: Control

SUMMARY:
Americans only receive 50% of indicated preventive services. We hypothesize that an interactive preventive health record (IPHR) will increase the delivery of recommended screening tests, immunizations, and counseling. The IPHR will function as a highly sophisticated personal health record for prevention, linking patients directly to their health information in the electronic record of their primary care physician. The functions of the IPHR will extend beyond those of personal health records by providing tailored recommendations, links to educational resources and decision aids, and patient and clinician reminders. Year one will focus on updating and refining an existing IPHR prototype. The second and third year, through a randomized controlled trial, will examine the effectiveness of the IPHR. Outcomes will include (1) whether the IPHR increases the delivery of recommended preventive services, (2) whether participants use the IPHR, and (3) whether the IPHR increases shared decision-making and improves clinician-patient communication. The study will take place in seven primary care practices in the Virginia Ambulatory Care Outcomes Network (ACORN) that utilize a common electronic medical record (EMR). A randomly selected sample of 5,500 of the practices' 228,000 patients, stratified by age and gender, will be assigned in a one-to-one ratio to receive a request from their clinician to use the IPHR (intervention group) or receive "usual" preventive care (control group). A Preventive Services Survey, which uses standardized questions to evaluate the delivery of preventive care, will be mailed to 4,500 patients and the CAHPS Clinician & Group Survey will be mailed to 1,000 patients. Surveys will be mailed pre-intervention, 6 month post-intervention, and 18 months post-intervention. Delivery of preventive care will be measured by the Preventive Services Survey and EMR data, while shared decision-making and clinician-patient communication will be measured by the CAHPS survey. The change from baseline to 6 and 18 months post-intervention for the control and intervention groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients seen in the study practices within the previous year

Exclusion Criteria:

* Age <18 years
* Age >75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5500 (Actual)
Dates: Start 2007-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The proportion of control and intervention subjects who are current on EACH individual indicated preventive service | Annual for three years
The proportion of control and intervention subjects who are current on ALL indicated preventive services | Annual for three years
The mean score for intervention and control subjects for quality of clinician communication (CAPHS-CGS questions 14-20); and frequency with which patients report sharing medical decisions (CAHPS questions SD 1-3) | Annual for three years

SECONDARY OUTCOMES:
The proportion of intervention subjects who visit the IPHR and establish an account | During enrollment period

CONTACTS AND LOCATIONS:
Overall Officials: Alex H Krist, MD MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Fairfax Family Practice Centers, Fairfax, Virginia, United States

REFERENCES:
- [Background] Krist AH, Peele E, Woolf SH, Rothemich SF, Loomis JF, Longo DR, Kuzel AJ. Designing a patient-centered personal health record to promote preventive care. BMC Med Inform Decis Mak. 2011 Nov 24;11:73. doi: 10.1186/1472-6947-11-73. PMID 22115059
- [Background] Krist AH, Woolf SH. A vision for patient-centered health information systems. JAMA. 2011 Jan 19;305(3):300-1. doi: 10.1001/jama.2010.2011. No abstract available. PMID 21245186
- [Result] Krist AH, Woolf SH, Rothemich SF, Johnson RE, Peele JE, Cunningham TD, Longo DR, Bello GA, Matzke GR. Interactive preventive health record to enhance delivery of recommended care: a randomized trial. Ann Fam Med. 2012 Jul-Aug;10(4):312-9. doi: 10.1370/afm.1383. PMID 22778119
- [Derived] Kerns JW, Krist AH, Longo DR, Kuzel AJ, Woolf SH. How patients want to engage with their personal health record: a qualitative study. BMJ Open. 2013 Jul 30;3(7):e002931. doi: 10.1136/bmjopen-2013-002931. PMID 23901027
- See also: A How-To Guide for Using Patient-Centered Personal Health Records to Promote Prevention — http://healthit.ahrq.gov/KRIST-IPHR-Guide-0612.pdf